CLINICAL TRIAL: NCT07331623
Title: Comparative Effects of Moderate Intensity Circuit Training and Moderate-Intensity Continuous Training on Heart Rate Recovery, VO2 Max, Power and Agility in Soccer Players
Brief Title: Comparative Effects of Moderate Intensity Circuit Training and Moderate-Intensity Continuous Training in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0476
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Moderate intensity Circuit Training; Moderate-Intensity Continuous Training; Soccer players

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (MICT) (Experimental): Group A was administered Moderate-intensity continuous Training protocol along with the baseline warm-up regime
  Interventions: Other: Moderate-intensity continuous Training
- Group B (MICT-CT) (Experimental): Group B was administered Moderate-intensity circuit training protocol along with the baseline warm-up regime.
  Interventions: Other: Moderate-Intensity Circuit Training

INTERVENTIONS:
Other: Moderate-intensity continuous Training — Group A: Experimental Group (MICT)
  Frequency: 2 times/week Duration: 45 minutes/session
  Structure:
  Warm-Up (10 minutes): Stationary Marching, Toe Touches, Leg/Arm Swings, Rotations, Push-Ups, Lunges, Bodyweight Squats.
  Primary Exercise (25 minutes):
  MICT Protocol: 8 sets of 4 minutes each (20s all-out effort, 10s rest) at 60-70% of HRmax.
  Exercises: Forward Lunges, Jump Squats, Burpees, Spider Crawls, Planks, Mountain Climbers, Ab Crunches. (At moderate intensity and controlled pace) Cool-Down (10 minutes): Static Stretching (Hamstring, Quad, Shoulder, Child's Pose).
  Arms: Group A (MICT)
Other: Moderate-Intensity Circuit Training — Group B: Contrast Group (Circuit Training of Moderate intensity)
  Frequency: 2 times/week Duration: 45 minutes/session
  Structure:
  Warm-Up (10 minutes): Same as Group A.
  Primary Exercise (25 minutes):
  Circuit: 30s per exercise, 15s rest, 3 sets with 45s rest between sets. Exercises: Jump Rope, Butterfly Sit-Ups, Hurdle Hop, Push-Ups, Jack-Knife, Squats, Inverse Sit-Ups.
  Cool-Down (10 minutes): Same as Group A.
  Arms: Group B (MICT-CT)

SUMMARY:
This study will compare the effects of Moderate-Intensity Circuit Training (MICT) and Moderate-Intensity Continuous Training (MICT) on Heart rate recovery, VO₂ max, power, and agility in 40 male soccer players aged 18-25. Participants will be randomly assigned to either group, with two 45-minute sessions per week over 8 weeks. Pre- and post-intervention assessments will include heart rate recovery, VO₂ max, 5 Jump Test, and T-Test for agility. Statistical analyses will compare within- and between-group changes using paired t-tests and ANOVA. The goal is to determine which training method is more effective for enhancing athletic performance.

DETAILED DESCRIPTION:
Study design: Randomized clinical trial Sample Size: To be calculated

Inclusion Criteria:

* Male soccer players aged 18-35 years.
* Players with at least two years of competitive soccer experience and are in practice season.
* Players with a body mass index (BMI) within the range of 18.5 to 30 kg/m².
* Availability to attend all training sessions and assessments.

Exclusion Criteria:

* Participants with medical conditions that contraindicate exercise.
* Athletes currently involved in other Moderate-Intensity continuous training programs.
* Presence of cardiovascular, neuromuscular, orthopedic, or neurologic conditions.
* Individuals who have undergone any surgery in the past six months.
* Those who do not provide written informed consent.
* Players taking any nutritional supplements, drugs, nicotine and alcohol.
* Athletes with known sleep disorders.

Sampling Technique:

Non probability purposive sampling technique.

Tools:

1. Heart Rate Recovery (HRR) Assessment
2. VO2 Max - Multistage Fitness Test (MSFT)
3. Power Assessment: 5 Jump Test
4. Agility Assessment: T-Test

ELIGIBILITY:
Inclusion Criteria:

* Male soccer players aged 18-35 years.
* Players with at least two years of competitive soccer experience and are in practice season.
* Players with a body mass index (BMI) within the range of 18.5 to 30 kg/m².
* Availability to attend all training sessions and assessments

Exclusion Criteria:

* Participants with medical conditions that contraindicate exercise.
* Athletes currently involved in other Moderate-Intensity continuous training programs.
* Presence of cardiovascular, neuromuscular, orthopedic, or neurologic conditions.
* Individuals who have undergone any surgery in the past six months.
* Those who do not provide written informed consent.
* Players taking any nutritional supplements, drugs, nicotine and alcohol.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Heart Rate Recovery | 8 weeks
  Heart Rate Recovery (HRR) measures how quickly the heart rate decreases after exercise, reflecting cardiovascular efficiency. Participants perform a 5-minute warm-up followed by a 3-minute step test using a 16.25-inch bench at a pace of 96 beats per minute. After completing the test, participants stand still, and heart rate is measured at the carotid pulse exactly 60 seconds post-exercise using a pulse oximeter. HRR is calculated as the difference between peak heart rate during exercise and heart rate after one minute. This test is used to assess cardiovascular recovery responses in soccer players following different training methods.
VO2 Max - Multistage Fitness Test (MSFT) | 8 weeks
  VO₂max represents aerobic capacity and overall cardiovascular fitness. It is estimated using the Multistage Fitness Test conducted on a 20-meter shuttle course. Participants run back and forth between two markers, starting at 8.5 km/h, with speed increasing by 0.5 km/h each minute, guided by audio beeps. The test ends when participants can no longer maintain the required pace. VO₂max is calculated using a standardized formula based on total running time, age, and number of shuttles completed, allowing comparison of aerobic capacity between training groups.
Power Assessment: 5 Jump Test | 8 weeks
  The 5 Jump Test assesses lower-body explosive power. Athletes begin behind a starting line and perform five continuous forward jumps, landing on both feet and immediately rebounding into the next jump without pausing. The total distance covered from the starting line to the final landing point is measured in centimeters. Adequate rest is provided between trials to ensure consistency. This test evaluates lower-limb power, which is essential for soccer performance.
4. Agility Assessment: T-Test | 8 weeks
  The T-Test measures agility by assessing rapid acceleration, deceleration, and directional changes. Cones are set in a T-shaped layout, with participants sprinting forward, shuffling laterally to both sides, and sprinting back to the start. Time is recorded from the initial movement to crossing the finish line. Lower completion times indicate better agility. This test is widely used to evaluate movement efficiency in soccer players.

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Hameed, MS SPT, Principal Investigator — Riphah International University; Maham Riaz, DPT, Principal Investigator — Riphah International University
Locations (1):
- Model Town Sports club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinho DV, Field A, Rebelo A, Gouveia ER, Sarmento H. A Systematic Review of the Physical, Physiological, Nutritional and Anthropometric Profiles of Soccer Referees. Sports Med Open. 2023 Aug 10;9(1):72. doi: 10.1186/s40798-023-00610-7. PMID 37561241
- [Background] Ramos-Campo DJ, Andreu Caravaca L, Martinez-Rodriguez A, Rubio-Arias JA. Effects of Resistance Circuit-Based Training on Body Composition, Strength and Cardiorespiratory Fitness: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Apr 28;10(5):377. doi: 10.3390/biology10050377. PMID 33924785
- [Background] Atakan MM, Li Y, Kosar SN, Turnagol HH, Yan X. Evidence-Based Effects of High-Intensity Interval Training on Exercise Capacity and Health: A Review with Historical Perspective. Int J Environ Res Public Health. 2021 Jul 5;18(13):7201. doi: 10.3390/ijerph18137201. PMID 34281138
- [Background] Fang B, Kim Y, Choi M. Effect of Cycle-Based High-Intensity Interval Training and Moderate to Moderate-Intensity Continuous Training in Adolescent Soccer Players. Healthcare (Basel). 2021 Nov 25;9(12):1628. doi: 10.3390/healthcare9121628. PMID 34946354
- [Background] McQuilliam SJ, Clark DR, Erskine RM, Brownlee TE. Effect of High-Intensity vs. Moderate-Intensity Resistance Training on Strength, Power, and Muscle Soreness in Male Academy Soccer Players. J Strength Cond Res. 2023 Jun 1;37(6):1250-1258. doi: 10.1519/JSC.0000000000004387. Epub 2023 Jan 18. PMID 36662035